CLINICAL TRIAL: NCT05004506
Title: A Prospective Randomized Controlled Trial of Intra-articular Analgesia Versus Adductor Canal Block for Arthroscopic Knee Surgery
Brief Title: Intra-articular Analgesia Versus Adductor Canal Block for Arthroscopic Knee Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Loyola University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LU208664
Record Dates: First submitted 2021-08-11; First posted 2021-08-13 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Post-Operative Pain, Chronic
MeSH Terms: conditions — Pain, Postoperative | interventions — Injections, Intra-Articular

STUDY DESIGN:
Intervention Model Description: Group A will be for single shot adductor canal block. Group B will receive the intra-articular injection.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): Group A patients will receive their treatment at the completion of the case while under general anesthesia. The anesthesia provider will identify the adductor canal using ultrasound guidance and inject 15ccs of 0.5% marcaine with epinephrine around the saphenous nerve.
  Group A patients will receive placebo intra-articular and arthroscopic portal site saline injections equal in volume and procedure time point as the treatment in Group B.
  At the completion of the case, the patient will be extubated and transferred to the PACU.
  Interventions: Drug: Adductor Canal Block
- Group B (Active Comparator): Group B will receive 20ccs of 2% lidocaine with epinephrine as an intra-articular injection. At the completion of the arthroscopic procedure the patient will receive an additional 20ccs of 0.5% marcaine with epinephrine intra-articular injection.
  Group B patients will also receive 10ccs of 2% lidocaine with epinephrine injected superficially into each of the arthroscopic portal sites. Group B patients will receive a 15cc saline injection around the saphenous nerve under the same procedure as the adductor canal block for Group A.
  At the completion of the case, the patient will be extubated and transferred to the PACU.
  Interventions: Drug: Intra-articular Injection

INTERVENTIONS:
Drug: Adductor Canal Block — The anesthesia provider will identify the adductor canal using ultrasound guidance and inject 15ccs of 0.5% marcaine with epinephrine around the saphenous nerve.
  Arms: Group A
Drug: Intra-articular Injection — receive 20ccs of 2% lidocaine with epinephrine as an intra-articular injection
  Arms: Group B

SUMMARY:
This study is a randomized study that compares two commonly used post-operative pain reducing techniques by measuring the level of pain and use of pain medication after knee surgery.

DETAILED DESCRIPTION:
Post-operative pain is a commonly associated with knee surgery. Treatment often includes an oral or intravenous (IV) narcotic regimen which often leads to nausea, vomiting and can cause consti-pation. These issues can contribute to the overall discomfort of the post-operative patient. Intra-operative injections and local nerve blocks have become common adjuncts to narcotics to reduce post-operative pain and the necessity for oral or IV narcotic use. The aim of this study is to com-pare analgesic use and clinical effects on post-operative pain management with intra-articular in-jection of 20ccs of 2% lidocaine with epinephrine at the start of the case plus 20ccs 0.5% mar-caine with epinephrine at the end of the case vs. adductor canal saphenous nerve blockade in pa-tients undergoing knee arthroscopy, as indicated by the need for rescue narcotics and patient pain scores. A randomized, single blinded study will be performed to evaluate post-operative pain control using VAS scores at 1, 2, 4, 8, 12, 24, 36, and 48hrs post-operatively, rescue narcotic use in the PACU, and total narcotic consumption over the same time period.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients
* Age 18 to 65 years

Exclusion Criteria:

* Allergy or intolerance to local anesthetics, NSAIDs, or opioids
* Inability to understand the consent or study process
* Any contraindication to regional anesthesia
* Known history of substance abuse
* Chronic home opioid therapy
* History of major neurologic deficit in operative limb
* Chronic pain syndromes
* Pregnancy and nursing women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04-20; Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Analgesic efficacy | 1, 2, 4, 8, 12, 24, 36, and 48 hours after surgery
  VAS pain scores
Rescue narcotics use | During post-surgical hospitalization
  Opioid requirement due to pain
Total narcotic consumption | During post-surgical hospitalization
  Opioid requirement overall

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No